CLINICAL TRIAL: NCT05756699
Title: A Prospective Study Evaluating the Accuracy of Proteome Multimarker Panel With Multiple Reaction Monitoring vs. Ultrasonography and Serum AFP as a Surveillance for Hepatocellular Carcinoma in High-Risk Population
Brief Title: Evaluation of Proteome Multimarker Panel With Multiple Reaction Monitoring as a Surveillance for Hepatocellular Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeong-Hoon Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH 2301-011-1391
Record Dates: First submitted 2023-02-20; First posted 2023-03-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After obtaining informed consent, a total of 40 cc of blood will be obtained from patients (20 cc x 2 times).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: multiple reaction monitoring (MRM)-based multimarker panel — multiple reaction monitoring (MRM)-based multimarker panel test to detect hepatocellular carcinoma

SUMMARY:
Most current guidelines recommend hepatocellular carcinoma (HCC) surveillance with ultrasound and alpha feto-protein (AFP) every 6 months for individuals with risk factors. However, the sensitivity of ultrasound for HCC detection is significantly reduced, especially in high-risk cirrhotic patients. In this study, the investigators aim to evaluate the efficacy of multiple reaction monitoring (MRM)-based multimarker panel as a surveillance tool for HCC. During two surveillance periods (starting from the time of voluntary consent and 6 months later), participants receive ultrasound, AFP, and MRM-based multimarker panel analysis. Patients who are suspected of HCC based on one of three tests undergo a contrast-enhanced CT scan within 6 weeks. After 6 months from the second surveillance period, the investigators re-evaluate the development of HCC using contrast-enhanced CT and AFP. The diagnostic accuracy of MRM-based multimarker panel is compared to ultrasound and AFP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis aged over 18 years, who receive regular surveillance for hepatocellular carcinoma.
* Patients with Risk Index greater than 2.33, corresponding to the annual 5% risk of hepatocellular carcinoma development.

  * Risk Index = 1.65 (if the prothrombin activity was ≤ 75%) + 1.41 (if the age was 55 years or older) + 0.92 (if the platelet count was < 75 X103/mm3) + 0.74 (if the presence of anti-hepatitis C virus was positive).

Exclusion Criteria:

* History of malignancy diagnosis including hepatocellular carcinoma
* Impaired renal function (Estimated glomerular filtration rate <30 mL/min/1.73m2)
* Impaired hepatic function (Child-Pugh class C)
* Patients who are not eligible for voluntary consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis who receive regular surveillance for hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HCC detection rate | Up to 2 years
  HCC detection using each surveillance modality/Total HCC cases

SECONDARY OUTCOMES:
Early HCC detection rate | Up to 2 years
  Early HCC (BCLC stage 0 or 1) detection using each surveillance modality/Total early HCC cases
False referral rate | Up to 2 years
  False-positive case of each surveillance modality/Total false-positive and false-negative results
Positive predictive value | Up to 2 years
  True-positive case of each surveillance modality/Total positive cases

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided